CLINICAL TRIAL: NCT02423291
Title: A Phase II Study of SGN-35 (Brentuximab Vedotin) of Patients With Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (PMLBCL)
Brief Title: A Study of SGN-35 (Brentuximab Vedotin) of Patients With Relapsed or Refractory PMLBCL
Acronym: FIL_SGN01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_SGN01
Record Dates: First submitted 2013-09-30; First posted 2015-04-22 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-04

CONDITIONS: Primary Mediastinal Large B Cell Lymphoma
Keywords: PMLBCL; Brentuximab Vedotin; CD30-positive; Mediastinal Lymphoma
MeSH Terms: interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vial for IV infusion (Experimental): This is a single-arm, open-label, multicenter, Phase 2 clinical trial to evaluate the efficacy and safety of Brentuximab vedotin as a single agent in patients with relapsed or refractory PMLBCL who have previously received a first line of treatment with chemotherapy or immunotherapy.20 patients will be treated in this study and All patients will receive 1.8 mg/kg Brentuximab vedotin administered as a single outpatient IV infusion on Day 1 of each 21-day treatment cycle. Patients may continue on study treatment until disease progression or unacceptable toxicity. Patients who achieve stable disease or better as assessed by investigator should receive a minimum of 8, but no more than 16 cycles of study treatment.
  Interventions: Drug: Brentuximab Vedotin

INTERVENTIONS:
Drug: Brentuximab Vedotin — Brentuximab vedotin, 1.8 mg/kg, administered via outpatient IV infusion on Day 1 of each 21-day cycle.
  Other Names: SGN-35; Adcetris

SUMMARY:
Study Objectives Primary:

• To determine the antitumor efficacy of single-agent Brentuximab vedotin (1.8 mg/kg administered intravenously every 3 weeks) as measured by the overall objective response rate in patients with relapsed or refractory primary mediastinal large B-cell lymphoma.

Secondary:

* To assess duration of tumor control, including duration of response and progression-free survival
* To assess survival
* To assess the safety and tolerability of Brentuximab vedotin

Additional:

• To assess disease-related symptoms

Number of Planned Patients 20 patients will be enrolled in this study. Duration of the study The study duration is 18 months for enrollment and 2 years for the follow-up.

DETAILED DESCRIPTION:
Study Population Eligible patients are those with relapsed or refractory primary mediastinal large B-cell lymphoma. Patients must also have histologically-confirmed CD30-positive disease, fluorodeoxyglucose (FDG)-avid and measurable disease of at least 1.5 cm, an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, and adequate hematologic, kidney, and liver function.

Eligible patients must not previously have been treated with Brentuximab vedotin or previously received an allotransplant. In addition, patients must not have congestive heart failure, known cerebral/meningeal disease, or any active viral, bacterial, or fungal infection requiring treatment with antimicrobial therapy within 2 weeks prior to first study dose.

Study Design This is a single-arm, open-label, multicenter, clinical trial to evaluate the efficacy and safety of Brentuximab vedotin as a single agent in patients with relapsed or refractory primary mediastinal large B-cell lymphoma.

Brentuximab vedotin will be administered as a single IV infusion on Day 1 of each 21-day cycle. Measures of anti-cancer activity will be assessed using the revised response criteria for malignant lymphoma. CT scans (chest, neck, abdomen, and pelvis) will be performed at baseline and Cycles 2, 4, 7, 10, 13, and 16 and PET scans will be done at baseline and Cycles 4 and 7. Patients will have an EOT assessment 30 ± 7 days after receiving their final dose of study drug. Long-term follow-up assessments (including survival and disease status information) will be performed every 12 weeks until either patient death or study closure, whichever occurs first. Patients who discontinue study treatment with stable disease or better will have CT scans done every 12 weeks until disease progression.

Test Product, Dose, and Mode of Administration Brentuximab vedotin, 1.8 mg/kg, administered via outpatient IV infusion on Day 1 of each 21-day cycle.

Number of Planned Patients 20 patients will be enrolled in this study. Duration of Treatment Brentuximab vedotin will be administered as a single IV infusion on Day 1 of each 21-day cycle. Patients may continue on study treatment until disease progression or unacceptable toxicity. Patients who achieve stable disease or better should receive a minimum of 8, but no more than 16 cycles of study treatment.

Duration of the study The study duration is 18 months for enrollment and 2 years for the follow-up. Efficacy Assessments Treatment response will be assessed by tumor imaging (spiral CT of neck, chest, abdomen, pelvis and PET scans) performed at protocol-specified timepoints. Determination of antitumor efficacy will be based on objective response assessments made according to the Revised Response Criteria for Malignant Lymphoma. Clinical response of progressive disease (PD), stable disease (SD), partial remission (PR), or complete remission (CR) will be determined at each assessment. Responses will be determined by investigator.

Safety Assessments Assessment of safety during the course of this study will consist of the surveillance and recording of adverse events (AEs), recording of concomitant medication and measurements of protocol-specified physical examination findings and laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for this study:

1. Patients with relapsed or refractory PMLBCL who have previously received at least 1 line of treatment. Patients must have completed any prior treatment with radiation, chemotherapy, biologics, immunotherapy and/or other investigational agents at least 4 weeks prior to the first dose of Brentuximab vedotin.
2. Histologically-confirmed CD30-positive disease.
3. Age greater than or equal to 18 years.
4. Fluorodeoxyglucose (FDG)-avid and measurable disease of at least 1.5 cm as documented by both PET and spiral CT.
5. An Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. The following required baseline laboratory data: absolute neutrophil count (ANC) ≥1500/μL, unless known marrow involvement due to disease, platelets ≥75,000/μL, unless known marrow involvement due to disease, bilirubin ≤1.5X upper limit of normal (ULN) or ≤3X ULN for patients with Gilbert's disease, serum creatinine ≤1.5X ULN, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5X ULN.
7. Serum Albumin ≥3 gr/dL;
8. Females of childbearing potential must have a negative serum or urine β-hCG pregnancy test result within 7 days prior to the first dose of Brentuximab vedotin. Females of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy.
9. Both females of childbearing potential and males who have partners of childbearing potential must agree to use two effective contraceptive methods during the study and for 30 days following the last dose of study drug.
10. Male patients, even if surgically sterilized (i.e., post vasectomy), who:

    * Agree to practice effective barrier contraception during the entire study treatment period and through 6 months after the last dose of the study drug, or
    * Agree to completely abstain from heterosexual intercourse
11. Patients or their legally authorized representative must provide written informed consent.

Exclusion Criteria:

1. Previous treatment with Brentuximab vedotin.
2. Previously received an allogeneic transplant.
3. Congestive heart failure, Class III or IV, by the NYHA criteria.
4. History of another primary malignancy for at least 3 years. (The following are exempt from the 3-year limit: nonmelanoma skin cancer, curatively treated localized prostate cancer, and cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on PAP smear.)
5. Known cerebral/meningeal disease.
6. Signs or symptoms of progressive multifocal leukoencephalopathy (PML).
7. Pre-existing Peripheral Neuropathy ≥ 2;
8. Any active systemic viral, bacterial, or fungal infection requiring treatment with antimicrobial therapy within 2 weeks prior to the first dose of Brentuximab vedotin.
9. Current therapy with other systemic anti-neoplastic or investigational agents.
10. Therapy with corticosteroids at greater than or equal to 20 mg/day prednisone equivalent within 1 week prior to the first dose of Brentuximab vedotin.
11. Women who are pregnant or lactating and breastfeeding.
12. Patients with a known hypersensitivity to recombinant proteins, murine proteins, or any excipient contained in the drug formulation.
13. Known human immunodeficiency virus (HIV) positive.
14. Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection.
15. Patients with dementia or an altered mental state that would preclude the understanding and rendering of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pier Luigi Zinzani, Prof., Principal Investigator — Istituto di Ematologia L. e A. Seragnoli - Bologna - Italy
Locations (9):
- Italy (9):
  - S.C. Ematologia A.O. SS. Antonio e Biagio e C. Arrigo, Alessandria, AL
  - Unità funzionale di Ematologia A.O.U. Careggi, Florence, FI
  - Dip. Oncologia, Ematologia e Patologie dell'apparato respiratorio A.O.U. Policlinico di Modena, Modena, MO
  - Divisione di Ematologia Azienda Ospedaliera "Bianchi Melacrino Morelli", Reggio Calabria, RC
  - S. C. Ematologia IRCCS Azienda Ospedaliera Arcispedale "S.Maria Nuova", Reggio Emilia, RE
  - Dipartimento di Biotecnologie Cellulari ed Ematologia Università "La Sapienza", Roma, Roma
  - S.C.D.O. Ematologia 2 A.O. Città della Salute e della Scienza, Torino, TO
  - Istituto di Ematologia L. & A. Seragnoli, Bologna
  - Ematologia Ospedale Businco, Cagliari

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vial for IV Infusion
Started | 15 (Patients enrolled)
Completed | 0 (Patients that have completed therapy)
Not Completed | 15
Not completed — Lack of Efficacy | 14
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vial for IV Infusion
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (18.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 15

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response Rate in Patients With Relapsed or Refractory PMLBCL
Description: The antitumor efficacy of single-agent Brentuximab vedotin (1.8 mg/kg administered intravenously every 3 weeks) as measured by the overall objective response rate in patients with relapsed or refractory primary mediastinal large B-cell lymphoma was determined using Cheson BD, Pfistner B, Juweid ME, et al. "Revised response criteria for malignant lymphoma". J Clin Oncol. 2007 Feb 10;25(5):579-586.Treatment response was assessed by dedicated spiral CT scan of neck, chest, neck, abdomen, and pelvis and PET scans performed at protocol-specified time points. Clinical response of progressive disease (PD), stable disease (SD), partial remission (PR), or complete remission (CR) will be determined at each assessment.
Time Frame: 42 months
Population: Trial was closed due to drug inefficacy on 14/Jul/2016 (last enrollment on 30/Jun/2015). Details in the Outcome Measure Data Table.
Measure: Count of Participants; unit: Participants
Arm/Group | Vial for IV Infusion
Number analyzed (Participants) | 15
Participants
  Quick PD | 11
  PD after 1 cycle | 1
  PD after 2 cycle | 1
  PR | 1
  SAE not related to drug | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected durig all Study Duration (3 years, 10 months).
Description: We used the Common Terminology Criteria for Adverse Events v. 4.0 (CTCAE) for the coding of adverse events.
Arm/Group | Vial for IV Infusion
All-Cause Mortality (participants affected / at risk) | 3/15
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vial for IV Infusion (N=15)
Tachycardia (Cardiac disorders) | 1 (1) — CARDIAC DISORDER Tachycardia
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vial for IV Infusion (N=15)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Peripheral neuropathy (NEC) (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Granulocytopenia (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No